CLINICAL TRIAL: NCT06577636
Title: Efficacy of Anesthesia-induced Dreaming for Post-traumatic Stress Disorder: a Randomized Controlled Trial
Brief Title: Induction of Dreaming With EEG and Anesthesia for Post-traumatic Stress Disorder
Acronym: IDEA_PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Boris D. Heifets, Associate Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 76919
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Post-traumatic Stress Disorder
Keywords: anesthesia; propofol; PTSD; post-traumatic stress disorder; dreaming; dreams
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Two groups of participants will be randomized to either (a) Dream experiences group, or (b) Non-Dream experiences group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham-controlled RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dream Experiences Group (Experimental): This group (n=21) will be subjected to an emergence-from-loss of responsiveness (LOR) protocol intended to elicit dream reports.
  Interventions: Procedure: Propofol anesthesia
- Non-Dream Experiences Group (Sham Comparator): This Group (n=21) will be subjected to a light sedation without loss of responsiveness protocol, designed to elicit non-dream experiential reports while responsive.
  Interventions: Procedure: Propofol anesthesia
- Open-label anesthesia protocol (Experimental): All participants (n = 15) will be subjected to an emergence-from-loss of responsiveness (LOR) protocol intended to elicit dream reports AND to a light sedation without loss of responsiveness protocol intended to elicit non-dream experiential reports while responsive.
  Interventions: Procedure: Propofol anesthesia

INTERVENTIONS:
Procedure: Propofol anesthesia — EEG-guided infusion of anesthestetics

SUMMARY:
The goal of this study is to test whether anesthesia-induced dreaming can help alleviate symptoms of PTSD in an (1) open-label trial (Phase I) and (2) double-blind, randomized controlled trial (Phase II) in a non-surgical setting. The investigators predict that inducing and sustaining a dream state prior to emergence from anesthesia will result in reduced symptoms of PTSD. Participants will undergo EEG-guided propofol anesthesia during which they will be either (1) receiving deep sedation leading to loss of responsiveness, designed to elicit dream reports upon emergence (Dream Protocol), and/or (2) light sedation without loss of responsiveness, designed to elicit non-dream experiential reports while responsive (e.g., simple imagery, sounds, thoughts, bodily sensations, hypnagogic-like experiences) (Non-Dream Protocol). The investigators will then investigate whether the deep-sedation Dream Condition is associated with a larger reduction in PTSD symptoms than the light-sedation Non-Dream Condition.

DETAILED DESCRIPTION:
GENERAL BACKGROUND

Post-traumatic stress disorder (PTSD) affects millions of Americans, and it can make everyday life very challenging. PTSD is characterized by recurrent distressing memories and nightmares, flashbacks, hyperarousal, and avoidance of things that remind individuals of their traumatic event. Nightmares reflect impaired emotion regulation occurring during sleep. There is evidence that therapeutic applications of dreaming may help target nightmares and other PTSD symptoms because dreaming is involved in memory (re)processing and emotion regulation. There is preliminary evidence that dreaming during anesthesia may reduce symptoms of PTSD. However, larger studies are needed to systematically test this.

AIM AND HYPOTHESES

The aim of this study is to test the efficacy of anesthesia-induced dreaming for PTSD in a (1) open-label trial (Phase I) and (2) double-blind, randomized controlled trial (Phase II) in a non-surgical setting. The investigators predict that inducing and sustaining a dream state prior to emergence from anesthesia will result in reduced symptoms of PTSD.

STUDY DESIGN

Design:

Phase I : Open-label study Phase II: Double-blind, sham-controlled RCT

Sample Size:

Phase I: N = 15 Phase II: N = 42 (21 in Dream Condition, 21 in Non-Dream Condition)

Variables:

Phase I and II: Outcome variables include: (1) Clinician-Administered PTSD Scale for DSM-5 (CAPS-5); (2) PTSD Checklist for DSM-5 (PCL-5)

STUDY PROCEDURES AND MEASURES

This research study is expected to take approximately 3 months to complete (per participant). During this time, participants will make 1 screening visit via zoom and 1 in-person screening visit at Stanford Hospital. Participants will also complete daily assessments of sleep quality and dream experiences 2 weeks before and 2 weeks after the anesthesia session. In Phase I, participants will also wear the Muse headband to measure sleep quantity and quality daily for 2 weeks before and 2 weeks after the intervention session. Participants will fill in pre-anesthesia and post-anesthesia questionnaires measuring mental health and well-being and, complete follow-up measures 1 week, 2 weeks, 1 month, and 3 months after the anesthesia session.

During the anesthesia session, participants will undergo EEG-guided infusion of propofol.

In Phase I, all participants will undergo at least two sessions: (1) an emergence-from-loss of responsiveness (LOR) protocol intended to elicit dream reports (Dream Condition); and (ii) light sedation without loss of responsiveness, designed to elicit non-dream experiential reports while responsive (e.g., simple imagery, sounds, thoughts, bodily sensations, hypnagogic-like experiences) (Non-Dream Condition).

In Phase II, participants will be randomized into either the Dream or Non-Dream Group, undergoing either the protocol designed to elicit dream experiences or non-dream experiences during no-LOR, respectively.

Immediately upon emerging from anesthesia, participants will be interviewed using the modified Brice questionnaire and their responses audio recorded.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion when all of the following criteria are met:

1. Male or female, 18 to 70 years of age
2. Able to read, understand, and provide written, dated informed consent prior to screening.
3. Diagnosed with PTSD prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition. The diagnosis of PTSD will be made by a trained study staff member and supported by the Structured Clinical Interview for DSM Disorders (SCID).
4. Meet the threshold of CAPS-5 score of >20 during screening.
5. In sufficiently good health to proceed with a low-risk elective procedure, characterized using the American Society of Anesthesiologists (ASA) physical status classification system as Class I or II.
6. If female, a status of non-childbearing potential or use of an acceptable form of birth control
7. Body mass index between 17-35 kg/m2.

Exclusion Criteria:

A potential participant will NOT be eligible for participation if any of the following criteria are met:

1. Female who is pregnant or breastfeeding.
2. Total CAPS-5 score ≤20 at either the screening.
3. Current diagnosis of a Substance Use Disorder (SUD; Abuse or Dependence, as defined by DSM-V) rated "moderate" or "severe" per criteria of the SCID, or Alcohol Use Disorder rated "moderate" or "severe" per SCID criteria. The following categories of SUD will NOT be excluded: nicotine dependence; alcohol or substance use disorder rated "mild"; alcohol or substance use disorder of any severity in remission, either early (3-12 months) or sustained (>12 months) time frames.
4. Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Specific Phobia, or Bipolar II Disorder (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more)
5. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
6. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within five years of screening.
7. Any Axis I or Axis II Disorder, which at screening is clinically predominant to their PTSD or has been predominant to their PTSD at any time within six months prior to screening.
8. In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of his/her participation in the study.
9. A neurological disorder
10. A cardiovascular disorder
11. A pulmonary/respiratory disorder
12. Clinically significant liver disease
13. Clinically significant kidney disease
14. Symptomatic gastroesophageal reflux disease, hiatal hernia, or other gastrointestinal disorder placing patient at risk for aspiration or that would merit categorization of patient as ASA Class III or higher
15. An endocrine disorder
16. Any other abnormal laboratory result at the time of the screening exam that in the view of the investigator poses a risk for participation in the study.
17. If, in the view of the participant's current primary mental health care provider this study poses a risk for participation (if a participant has a current mental health care provider).
18. Participation in any clinical trial with an investigational drug or device that conflicts with this trial, within the past month or concurrent to study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | 1 month post-intervention
  The CAPS-5 is a structured interview that is considered the gold standard for assessing post-traumatic stress disorder (PTSD). The CAPS-5 is designed to assess the 20 symptoms of PTSD as defined by the DSM-5, as well as the impact of these symptoms on social and occupational functioning. The CAPS-5 includes 20 items corresponding to the DSM-5 criteria for PTSD. Each item is rated for both frequency and intensity, with a 5-point scale (0-4) for each dimension. The total score ranges from 0 to 80, with higher scores indicating more severe symptoms. A score of >20 points indicates clinically significant PTSD symptoms. Superiority of "Dream Experiences Group" over "Non-Dream Experiences Group" will be demonstrated by a statistically significant greater decrease in the CAPS-5 when comparing pre-anesthesia scores to post-anesthesia scores.

SECONDARY OUTCOMES:
Number of Participants With Clinical Response | 1 month post-intervention
  Clinical response is defined as a reduction of ≥15 points (or ≥30% - 50%) in the score of CAPS-5 in the Dream Experiences Group, comparing baseline pre-anesthesia scores to post-anesthesia scores.
Number of Participants With Remission | 1 month post-intervention
  Remission is defined as obtaining a score of ≤20 points on the CAPS-5 in the Dream Experiences Group post-intervention.
PTSD Checklist for DSM-5 (PCL-5) | 1 month post-intervention
  The PCL-5 is a self-report measure designed to assess the 20 symptoms of post-traumatic stress disorder (PTSD) as defined by the DSM-5. Includes 20 items that correspond directly to the DSM-5 criteria for PTSD. Each item is rated on a 5-point Likert scale from 0 (Not at all) to 4 (Extremely), indicating how much the symptom has bothered the individual in the past week/month. The total score can range from 0 to 80, with higher scores indicating more severe PTSD symptoms. A score of 31-33 or higher is considered indicative of symptomatic PTSD. Superiority of the Dream vs No-Dream group will be demonstrated by a reduction of ≥30% - 50% in the self-reported PTSD symptoms, as measured with the PCL-5, comparing baseline pre-anesthesia scores to post-anesthesia scores.

CONTACTS AND LOCATIONS:
Overall Officials: Boris D Heifets, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiers might be removed from identifiable private information and/or identifiable specimens and, after such removal, the information and/or specimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from the participant.
  The results of this research study may be presented at scientific or medical meetings or published in scientific journals without disclosing the identify of the participants (unless there is a separate consent from participants to reveal their identity).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available after the results of the study have been analyzed and published
Access Criteria: We will share the information via Open Science Framework (osf.io), github, or via official Stanford file sharing options

REFERENCES:
- [Background] Hack LM, Sikka P, Zhou K, Kawai M, Chow HS, Heifets B. Reduction in Trauma-Related Symptoms After Anesthetic-Induced Intra-Operative Dreaming. Am J Psychiatry. 2024 Jun 1;181(6):563-564. doi: 10.1176/appi.ajp.20230698. Epub 2024 Mar 13. No abstract available. PMID 38476046
- [Background] Chow HS, Hack LM, Kawai M, Heifets BD. Anesthetic-Induced Intraoperative Dream Associated With Remission of a Psychiatric Disorder: A Case Report. A A Pract. 2022 Aug 10;16(8):e01613. doi: 10.1213/XAA.0000000000001613. eCollection 2022 Aug 1. PMID 35952341
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729